CLINICAL TRIAL: NCT07056348
Title: Chronic Stimulation of the Motor Ventral Thalamus (VOP/VIM) for Motor Control in Humans
Brief Title: Long-term Brain Stimulation of the Motor Ventral Thalamus (VOP/VIM) to Improve Motor Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Gonzalez-Martinez (Other)
Responsible Party: Sponsor-Investigator, Jorge Gonzalez-Martinez, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21100020
Record Dates: First submitted 2025-06-25; First posted 2025-07-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury; Stroke; Brain Disease; Movement Disorders (Incl Parkinsonism); Central Nervous System Disease; Essential Tremor, Movement Disorders; Essential Tremor of Voice
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Brain Diseases; Movement Disorders; Central Nervous System Diseases; Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open-label, descriptive, experimental.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Deep Brain Stimulation of the Motor Thalamus (Experimental): Individuals with deep brain stimulation device implanted in the motor thalamus for movement disorders treatment who also sustain speech, swallowing, and motor deficits.
  Interventions: Device: Deep Brain Stimulation (DBS) of the Motor Thalamus
- Healthy Control Participants (No Intervention): The investigators aim to include healthy control subjects who will complete the language and upper-limb tasks. The healthy subjects will not undergo any surgical procedures.

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) of the Motor Thalamus — All participants enrolled will undergo stimulation parameters tuning of deep brain stimulation electrode leads. All subjects will participate in a series of experiments to evaluate the stimulation effects on movement of face and upper extremities, swallowing, and speech abilities.
  Arms: Deep Brain Stimulation of the Motor Thalamus

SUMMARY:
This study aims to recruit patients already implanted with Deep Brain Stimulation (DBS) for movement disorders to complete tasks assessing parameters of motor output, speech, and swallowing functions, both with and without stimulation. DBS parameters would be adjusted prior to motor testing. Patients would then participate in multiple sessions performing contralateral upper extremity movement tasks measuring movement speed, grip strength, and strength modulation, facial movement, swallowing, and speech tasks.

DETAILED DESCRIPTION:
The study is designed to assess the assistive effects of DBS (i.e., immediate effects when the stimulation is turned ON) and obtain preliminary evidence for therapeutic effects (i.e., long-lasting effects with stimulation OFF). Researchers will 1) quantify the ability to recruit facial and oropharyngeal muscles with electrical stimulation of the motor thalamus in patients with DBS for movement disorders, 2) quantify the ability to recruit arm and hand muscles with electrical stimulation of the motor thalamus in patients with DBS, and 3) verify if the delivery of DBS has effects on the central nervous system with clinical measures.

ELIGIBILITY:
Inclusion Criteria:

* Movement disorder patients ≥18 years of age and < 80 years of age, who will be implanted with DBS for treatment of motor symptoms.
* Subject has provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, where applicable, prior to any study-related procedures.

Exclusion Criteria:

* History of seizure disorders
* Vasovagal response history and loss of consciousness history
* Severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator would impact participation in the study.
* Any serious disease or disorder (e.g. cancer, severe cardiac or respiratory disease, neurological conditions other than current movement disorder) or cognitive impairments that could impair ability to participate in this study.
* Females who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Motor Function - Hand Dexterity | 2 years
  The investigators will use the Box and Blocks Test (unit counts) and Brinkmann Test (unit counts) to measure hand dexterity. Based on the preliminary data, the investigators will consider the number of participants with an 18% change in hand dexterity as minimally acceptable for improvement. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Upper Limb Motor Function - Grip Strength | 2 years
  The investigators will use the Box and Blocks Test, Brinkmann Test, and force dynamometer tests to measure grip strength (Newton). These tests will combine weight and height into a single BMI measurement in kg/m^2. Based on the preliminary data, the investigators will consider the number of participants with an 18% change in grip strength as minimally acceptable for improvement. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Upper Limb Motor Function - Velocity | 2 years
  The investigators will use the Box and Blocks Test, Brinkmann Test, and force dynamometer tests to measure velocity (Newton per millisecond). These tests will combine weight and height into a single BMI measurement in kg/m^2. Based on the preliminary data, the investigators will consider the number of participants with an 18% change in velocity as minimally acceptable for improvement. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Upper Limb Motor Function - Strength Modulation | 2 years
  The investigators will use the Box and Blocks Test, Brinkmann Test, and force dynamometer tests to measure strength modulation (Newton). These tests will combine weight and height into a single BMI measurement in kg/m^2. Based on the preliminary data, the investigators will consider the number of participants with an 18% change in modulation as minimally acceptable for improvement. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Facial Muscle Motor Function | 2 years
  The investigators will use electromyography (EMG) testing to measure muscle strength and range of motion produced by the subject during isometric facial movements (e.g. smile, tongue out, puckered lips, and open-close mouth), measured in by calculation of Area-Under-the-Curve with units of uV^2/ms. These tests will combine weight and height into a single BMI measurement in kg/m^2. Based on the preliminary data, the investigators will consider the number of participants with an increase of 50% in ROM as a minimally acceptable improvement in muscle strength.
Swallowing Function | 2 years
  The investigators will use the modified barium swallow study (MBSS) to assess oropharyngeal swallow functions. This is a performance evaluation scale, that consist of 17 items with varying scales. The total score ranges from 0 to 55, where a higher score means a better outcome. Based on the preliminary data, the investigators will consider the number of participants with an increase of 1 point in at least 50% of the items of the Modified Barium Swallow Impairment Profile as a minimally acceptable improvement in swallow functions.
Speech Intelligibility | 2 years
  The investigators will use the Assessment of Intelligibility of Dysarthric Speech (AIDS) to assess the quality of communication and intelligibility of speech at both word- and sentence-level. Intelligibility is calculated as the percentage of words correctly identified in the single-word task, and as the percentage of correctly transcribed words and speech rate (in words per minute) in the sentence task. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 5% correctly transcribed to be minimally acceptable.
Dexterity of Articulation AMRs | 2 years
  The investigators will measure dexterity of articulation by alternating motion rates (AMRs) of the repetitive plosive sound (pah, tah, and kah). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Dexterity of Articulation SMRs | 2 years
  The investigators will measure dexterity of articulation by sequential motion rates (SMRs) of the repetitive plosive sound (pah, tah, and kah). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Oral Motor Functions | 2 years
  The investigators will use the 2nd Edition Frenchay Dysarthria Assessment (FDA-2) to measure patterns of oral motor functions, with a particular focus on the following subsections: Respiration, Lips, Palate, Laryngeal, and Tongue. Each subsection is rated on a scale from "a" to "e", where "a" means normal for age, and "e" means unable to undertake task/movement/sound. So a score closer to "a" means a better outcome. Based on the preliminary data, the investigators will consider the number of participants with an improvement in severity level (e.g., from considerable to moderate severity, or a score of D to C) to be minimally acceptable.
Respiration Capacity - Total Exhaled Volume | 2 years
  The investigators will measure pulmonary function and respiratory capacity by performing a spirometry test with focus on the forced vital capacity (FVC). The FVC is the total volume of air that can be forcefully exhaled after a maximal inhalation and this will be measured in liters (L). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 12% in the rate to be minimally acceptable.
Respiration Capacity - Volume Exhaled | 2 years
  The investigators will measure pulmonary function and respiratory capacity by performing a spirometry test with focus on the volume exhaled in the first second (FEV1). The FEV1 is the volume of air exhaled in the first second of a forced exhalation and this will be measured in liters (L). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 12% in the rate to be minimally acceptable.
Respiration Capacity - FEV1/FVC Ratio | 2 years
  The investigators will measure pulmonary function and respiratory capacity by performing a spirometry test with focus on ratio of the forced expiratory volume in one second (FEV1) to the forced vital capacity (FVC). The ratio is expressed as a unitless percentage. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 12% in the rate to be minimally acceptable.
Oral Motor Strength | 2 years
  The investigators will use the Iowa Performance Instrument (IOPI) to measure motor strength of tongue and lip using maximum force and endurance. IOPI instrument measures force applied from oral cavity by kPa. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gonzalez-Martinez, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 7 years from enrollment of the first participant.
Access Criteria: Data must be directly requested from the PI and will be shared upon completion of the necessary data-sharing agreement to protect confidential patient information.

REFERENCES:
- [Background] Franzini A, Cordella R, Nazzi V, Broggi G. Long-term chronic stimulation of internal capsule in poststroke pain and spasticity. Case report, long-term results and review of the literature. Stereotact Funct Neurosurg. 2008;86(3):179-83. doi: 10.1159/000120431. Epub 2008 Mar 12. PMID 18334861
- [Background] Phillips NI, Bhakta BB. Affect of deep brain stimulation on limb paresis after stroke. Lancet. 2000 Jul 15;356(9225):222-3. doi: 10.1016/s0140-6736(00)02487-9. PMID 10963204
- [Background] Cooper IS, Upton AR, Amin I. Reversibility of chronic neurologic deficits. Some effects of electrical stimulation of the thalamus and internal capsule in man. Appl Neurophysiol. 1980;43(3-5):244-58. doi: 10.1159/000102263. PMID 6975064
- [Background] Baker KB, Plow EB, Nagel S, Rosenfeldt AB, Gopalakrishnan R, Clark C, Wyant A, Schroedel M, Ozinga J 4th, Davidson S, Hogue O, Floden D, Chen J, Ford PJ, Sankary L, Huang X, Cunningham DA, DiFilippo FP, Hu B, Jones SE, Bethoux F, Wolf SL, Chae J, Machado AG. Cerebellar deep brain stimulation for chronic post-stroke motor rehabilitation: a phase I trial. Nat Med. 2023 Sep;29(9):2366-2374. doi: 10.1038/s41591-023-02507-0. Epub 2023 Aug 14. PMID 37580534
- [Background] Molnar GF, Sailer A, Gunraj CA, Cunic DI, Lang AE, Lozano AM, Moro E, Chen R. Changes in cortical excitability with thalamic deep brain stimulation. Neurology. 2005 Jun 14;64(11):1913-9. doi: 10.1212/01.WNL.0000163985.89444.DD. PMID 15955943
- [Background] Plow EB, Machado A. Invasive neurostimulation in stroke rehabilitation. Neurotherapeutics. 2014 Jul;11(3):572-82. doi: 10.1007/s13311-013-0245-y. PMID 24353109
- [Background] Lozano AM, Lipsman N, Bergman H, Brown P, Chabardes S, Chang JW, Matthews K, McIntyre CC, Schlaepfer TE, Schulder M, Temel Y, Volkmann J, Krauss JK. Deep brain stimulation: current challenges and future directions. Nat Rev Neurol. 2019 Mar;15(3):148-160. doi: 10.1038/s41582-018-0128-2. PMID 30683913
- [Background] Ho JC, Grigsby EM, Damiani A, Liang L, Balaguer JM, Kallakuri S, Tang LW, Barrios-Martinez J, Karapetyan V, Fields D, Gerszten PC, Hitchens TK, Constantine T, Adams GM, Crammond DJ, Capogrosso M, Gonzalez-Martinez JA, Pirondini E. Potentiation of cortico-spinal output via targeted electrical stimulation of the motor thalamus. Nat Commun. 2024 Oct 1;15(1):8461. doi: 10.1038/s41467-024-52477-1. PMID 39353911